CLINICAL TRIAL: NCT04592757
Title: Immersive Care - Virtual Mirror Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas More University of Applied Sciences (Other)
Collaborators: Revalidatieziekenhuis RevArte (Unknown); To Walk Again REVAlution Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC_REHAB_01
Record Dates: First submitted 2020-09-04; First posted 2020-10-19 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: Upper extremity; Rehabilitation; Virtual Reality; Immersive technology; Mirror therapy
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subacute stroke patients (Experimental): Training with new virtual mirror therapy application. During 12 sessions of approximately 30 minutes.
  Interventions: Device: Virtual mirror therapy via VR headset
- Chronic stroke patients (Experimental): Training with new virtual mirror therapy application. During 12 sessions of approximately 30 minutes.
  Interventions: Device: Virtual mirror therapy via VR headset

INTERVENTIONS:
Device: Virtual mirror therapy via VR headset — Participants will perform Activities of Daily Living (ADL) in a virtual environment through a VR headset. The application is based on mirror therapy. Participants will execute certain arm movements with their non-affected arm, while seeing their affected arm perform said movement in the virtual environment.
  Other Names: VR mirror therapy; VR application; Mirror therapy

SUMMARY:
The purpose of this implementation study is - primarily - to investigate the feasibility, acceptability, tolerability of a new virtual reality application in stroke patients, and -secondarily - to gain initial insights in the preliminary clinical effects of this application.

DETAILED DESCRIPTION:
Although immersive technologies have great potential in healthcare, they are still relatively unknown and underutilized in this field. In this study a new virtual reality (VR) application will be implemented and tested in two groups of stroke patients (10 acute phase/10 chronic phase). In an attempt to reactivate the affected upper limb in stroke patients, therapists often use mirror therapy. Using a mirror, the movement of a paralyzed limb is feigned in order to reprogram the brain. A patient performs exercises with the healthy limb, but through the mirror the patient seems to use the affected limb. A high number of repetitions is essential to stimulate the so-called neuroplasticity of the brain, but this makes mirror therapy monotonous. In addition, the therapy also has its limitations. Activities are limited by the physical boundaries of the modality, with exercises largely limited to distal movements and simple functional activities. Larger, free-standing mirrors provide a wider range of motion for therapeutic activities, but offer less protection against environmental distraction. With VR, these obstacles can be overcome. By focusing on virtual mirror therapy using a VR headset, therapists hope to create a more pleasant and realistic experience for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients in the subacute or chronic phase, aged between 18 and 85 years old with a normal functioning upper limb on the unaffected side and a reduced use and / or weakness and / or paralysis of the upper limb on the affected side
* Ability to sit on a chair or in a wheelchair with adequate trunk stability so that the unaffected upper limb can move freely
* Ability to follow verbal instructions
* Ability to communicate verbally with the researchers

Exclusion Criteria:

* Stroke patients in acute phase
* Severe medical conditions that interfere with the proper execution of the research
* Patients who are medically unstable
* Cognitive disorders which may complicate the research or make it impossible
* Speaking disorders (aphasia, dysarthria) which may complicate the proper execution of the research and the communication of important verbal information
* Visual disorders which complicate carrying out ADL activities or make it impossible
* Known allergies to any of the materials of the VR headset
* Epilepsy
* Extreme sensitivity to motion sickness
* Specific anxiety disorders that hinder the use of the VR headset such as claustrophobia
* Skin diseases or lesions in the contact area of the VR headset

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient attitude towards the VR mirror therapy | Before the start of the first session and immediately after finishing the last session.
  Assess change in patient attitude towards the VR mirror therapy with the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire survey. The UTAUT questionnaire survey for end-users consists of 20 items with five response options ranging from "Totally disagree" (1) to "Totally agree" (5), and returns scores ranging from 20 to 100. The questionnaire survey consists of 7 subscales, for most of which higher scores indicate a more positive attitude towards the VR mirror therapy.
Usability of the VR mirror therapy: System Usability Scale (SUS) | Immediately after finishing the last session.
  Assessment of ease of use of the VR mirror therapy with the System Usability Scale (SUS). The SUS is a 10-item questionnaire with five response options for respondents; from "strongly disagree" to "strongly agree", and returns scores ranging from 0 to 100. A higher SUS score indicates better usability.
Patient satisfaction: Client Satisfaction Questionnaire (CSQ-8) | Immediately after finishing the last session.
  Assessment of client satisfaction with the VR application with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 consists of 8 items with four response options and returns scores ranging from 8 to 32. Higher scores indicate higher satisfaction.
Therapy adherence | Immediately after finishing each session.
  Measure therapy adherence by registering the number of fully completed 30 min sessions.
Change from baseline in tolerability (Do participants experience symptoms of simulator sickness?) | Immediately after finishing the first and last session.
  Assessment of physical side effects after exposure to VR by the Simulator Sickness Questionnaire (SSQ).
Adverse event tracking | Up to 30 minutes during each session.
  Qualitative tracking of adverse events by patient observation scheme.

SECONDARY OUTCOMES:
Changes in pain levels from pre-to-post intervention session: Visual Analogue Scale | Immediately before and after each session.
  Assessment of changes in pain using a Visual Analogue Scale ranging from 0 = no pain at all, to 100 = most pain imaginable.
Change from baseline in functionality of the upper limb | Up to 10 minutes before the start of the first session and immediately after end of the last session.
  Assessment of changes in the functionality of the upper limb with the Fugl-Meyer upper extremity (FMUE) assessment. The FMUE Scale comprises 33 items, each scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully.

OTHER OUTCOMES:
Clinicians' assessment of usability: System Usability Scale (SUS) | After the last participant has finished the last session.
  Assessment of ease of use of the VR application with the System Usability Scale (SUS). The SUS is a 10 item questionnaire with five response options for respondents; from "strongly disagree" to "strongly agree", and returns scores ranging from 0 to 100. A higher SUS score indicates better usability.
Clinicians' satisfaction: Client Satisfaction Scale (CSQ-3) | After the last participant has finished the last session.
  Assessment of client satisfaction with the VR application with the Client Satisfaction Scale (CSQ-3). The CSQ-3 consists of 3 items with four response options and returns scores ranging from 3 to 12. Higher scores indicate higher satisfaction.
Clinicians' attitude towards VR mirror therapy | After the last participant has finished the last session.
  Assess clinicians' attitude towards technology with the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire. The UTAUT questionnaire survey for end-users consists of 31 items with five response options ranging from "Totally disagree" to "Totally agree", and returns scores ranging from 31 to 155. The questionnaire survey consists of 7 subscales, for most of which higher scores indicate a more positive attitude towards the VR mirror therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bernaerts, PhD, Principal Investigator — Thomas More University of Applied Sciences
Locations (2):
- Belgium (2):
  - Revalidatieziekenhuis RevArte, Edegem, Antwerpen
  - To Walk Again REVAlution Center, Herentals, Antwerpen

IPD SHARING:
Plan to Share IPD: No